CLINICAL TRIAL: NCT02098837
Title: An Open Label Study Examining the Efficacy and Cardiovascular Risk of Immediate Versus Deferred Switch From a Boosted PI to Dolutegravir (DTG) in HIV Infected Patients With Stable Virological Suppression
Brief Title: Cardiovascular Risk in HIV Patients Switching From a Boosted Protease Inhibitor (PI) to Dolutegravir (DTG)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEAT 22/SSAT 060
Record Dates: First submitted 2014-03-20; First posted 2014-03-28 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: HIV
Keywords: HIV
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate switch (Active Comparator): Patients will be randomised to switch from a boosted PI to dolutegravir at baseline.
  Interventions: Drug: Dolutegravir
- Deferred switch (Active Comparator): Patients will be randomised to switch from a boosted PI to dolutegravir after 48 weeks.
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir 50mg once daily
  Other Names: Tivicay

SUMMARY:
The purpose of the study is to investigate the benefits of switching away from a kind of drug called a boosted protease inhibitor (PI) to a new drug called dolutegravir on patients' cardiovascular health (the health of their hearts). Patients are currently taking two other anti-HIV drugs, called nucleoside reverse transcriptase inhibitors (NRTIs), with their boosted PIs; these NRTIs will not be changed throughout the study. In order to compare the boosted PI and dolutegravir more accurately, half of study participants will be switched to dolutegravir immediately, and the other half will be switched after 48 weeks of continuing on the boosted PI.

Boosted PIs are associated with increased heart and circulation risk so it is hoped that switching from a boosted PI to dolutegravir will improve the health of the patients' hearts. Dolutegravir is a drug for HIV treatment which has been approved for use in HIV patients in the US and Europe. Clinical trials using dolutegravir have found that it is effective at suppressing the HIV virus, and it is at least as effective as the other drugs.

This study will also investigate the safety (in terms of other side effects and the routine blood tests which the investigators ordinarily use to monitor patients' treatment) and monitor effectiveness, patients' viral load and CD4 counts, when patients switch treatment from a boosted PI to dolutegravir. Viral load is the amount of the HIV virus they have in their blood, and CD4 count is a measure of a type of cell that is in their immune system. We also aim to improve patients' cardiovascular health in general by providing them with information on how to live a healthy lifestyle (eg improving their diet, stopping smoking etc).

DETAILED DESCRIPTION:
Study Design: Randomised, non-inferiority strategic trial over 96 weeks with early or delayed switch from an ARV regimen containing a boosted PI plus 2 NRTIs to dolutegravir (DTG) plus 2 NRTIs in patients having achieved complete virological suppression for more than 24 weeks (HIV-1 RNA <50 c/ml). Patients will be randomised to switch at baseline or at 48 weeks.

Study visits will take place at screening, baseline, weeks 4 (immediate switch group only), 12, 24, 36, 48, 52 (deferred switch group only), 60, 72, 84 and 96, plus a follow up visit 28 days after the last dose of study medication.

Routine investigations will include viral load, CD4, haematology (including haemoglobin, white cell count and differential, platelets), biochemistry (including sodium, potassium, creatinine, albumin, glucose, ALT, ALP, total bilirubin, total cholesterol, HDL, LDL, triglycerides), quality of life questionnaires (EuroQL), urine sample (for haematuria, proteinuria, glycosuria, leukocytes, nitrate & pregnancy test in WOCBP)

ELIGIBILITY:
Inclusion Criteria:

* Patient volunteers who meet all of the following criteria are eligible for this trial:

  1. Is male or female aged over 50, OR aged over 18 years with a Framingham risk score above 10%
  2. Has documented HIV-1 infection
  3. Has signed the Informed Consent Form voluntarily
  4. Is willing to comply with the protocol requirements
  5. Has been receiving an ARV regimen containing a boosted PI (darunavir, atazanavir, lopinavir, or fosamprenavir) plus 2NRTIs for >24 weeks
  6. Has stable virological suppression (plasma HIV-RNA <50 copies/mL for >24 weeks)
  7. If female and of childbearing potential, is using effective birth control methods and is willing to continue practising these birth control methods during the trial and for at least 2 weeks after the last dose of study medication. Note: Non-childbearing potential is defined as either post-menopausal (12 months of spontaneous amenorrhoea and ≥45 years) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy
  8. If a heterosexually active male, he is using effective birth control methods and is willing to continue practising these birth control methods during the trial and until follow-up visit

Exclusion Criteria:

* Patients meeting 1 or more of the following criteria cannot be selected:

  1. Infected with HIV-2
  2. Using any concomitant therapy disallowed as per the reference safety information and product labelling for the study drugs
  3. Has acute viral hepatitis including, but not limited to, A, B, or C
  4. Has chronic hepatitis B and/or C with AST and/or ALT >5 x ULN Note: Subjects can enter trial with chronic HBV if HBV-DNA undetectable at screen (and no detectable result in last 6 months) and with chronic HCV if not expected to require treatment during the trial period.
  5. Any investigational drug within 30 days prior to the trial drug administration
  6. History of exposure to any ARVs other than PIs or NRTIs except if switch was for tolerability/toxicity (NOTE: patients who have previously taken part in single drug trials for less than 14 days need not be excluded, or for virological failure with a genotypic resistance test without mutations
  7. Any prior evidence of primary viral resistance based on the presence of any major resistance-associated mutation to backbone NRTI
  8. History of prior virological failure,eg 2 consecutive HIV-1 RNA >50 c/ml -at or after week 32 following first ART initiation or confirmed rebound viraemia >200 copies/ml after having a VL of <50 copies/ml without resistance test or with significant mutations to any other ARV regimen (NOTE: Switch for toxicity or tolerability with wild type virus does not count as virological failure)
  9. Dialysis or renal insufficiency (creatinine clearance < 50ml/min)
  10. History of decompensated liver disease (AST or ALT≥5x the upper limit of normal (ULN) or ALT ≥ )3 x ULN and bilirubin ≥ 1.5 x ULN with > 35% direct bilirubin.
  11. Unstable liver disease (as defined by the presence of ascities, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), know biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones))
  12. Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification
  13. If female, currently pregnant or breastfeeding
  14. Opportunistic infection within 4 weeks prior to first dose of DTG
  15. Clinical decision that a switch of antiretroviral therapy should be immediate
  16. Screening blood result with any grade 3/4 toxicity according to Division of AIDS (DAIDS) grading scale, except: asymptomatic grade 3 glucose, amylase or lipid elevation or asymptomatic grade 4 triglyceride elevation (re-test allowed).
  17. Any condition (including illicit drug use or alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the trial.
  18. History or presence of allergy to the study drug or their components

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2014-04; Primary Completion 2017-11 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Virological suppression | 48 weeks
  Maintenance of virological suppression (ie HIV-1 RNA <50 c/ml) after 48 weeks
Total cholesterol | 48 weeks
  Change from baseline in total cholesterol at week 48

SECONDARY OUTCOMES:
Virological Suppression | 24 - 96 weeks
  Maintenance of virological suppression (ie HIV-1 RNA <50 c/ml) at week 24 and 96
CD4 count from baseline | 24 - 96 weeks
  Change in CD4 count from baseline to week 24, 48 and 96
Baseline in total cholesterol | 24 - 96 weeks
  Change from baseline in total cholesterol at weeks 24 and 96
Change from baseline to lipid values | 24 - 96 weeks
  Change from baseline to lipid values (LDL, HDL, triglycerides and TC:HDL ratio) and Framingham and DAD scores at weeks 24, 48 and 96
Safety | 24 - 96 weeks
  Safety (clinical and laboratory adverse events) at weeks 24, 48 and 96
Changes in markers of inflammation | 48 - 96 weeks
  Changes in markers of inflammation at baseline, week 48 and week 96
Tolerability | 24 - 96 weeks
  Tolerability (EuroQoL questionnaire) at weeks 24, 48 and 96
Changes in markers of coagulation | 48 - 96 weeks
  Changes in markers of coagulation at baseline, week 48 and week 96
Changes in markers of endothelial dysfunction | 48 - 96 weeks
  Changes in markers of endothelial dysfunction at baseline, week 48 and week 96
Change to arterial stiffness augmentation index at weeks 48 and 96 | 48 - 96 weeks
  Change from baseline to arterial stiffness augmentation index at weeks 48 and 96
Change to average thickness of common carotid artery walls at weeks 48 and 96 | 48 - 96 weeks
  Change from baseline to average thickness of common carotid artery walls at weeks 48 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Jose Gatell, Dr, Principal Investigator — Spanish healthcare system
Locations (33):
- Belgium (3):
  - Insititute Of Tropical Medicine Antwerp, Antwerp
  - CHU Saint-Pierre, Brussels
  - Universitaire Ziekenhuis Gent, Ghent
- France (5):
  - Hopital de la Croix Rousse, Lyon
  - Service des Maladies Infectieuses et Tropicales du CHU de NANTES, Nantes
  - Hopital Saint Louis, Paris
  - Pitié-Salpêtrière Hospital, Paris
  - Hospital Bichat Claude-Bernard, Paris
- Germany (5):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Essen, Essen
  - Klinikum der Goethe-Universität Frankfurt, Frankfurt
  - ICH Infektiologisches Centrum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Italy (4):
  - Santa Maria Annunziata di Firenze, Florence
  - San Paolo Hospital, Milan
  - Azienda Ospedaliera - Polo Universitario 'Luigi Sacco', Milan
  - Universitaria di Modena, Modena
- Spain (8):
  - Universitario Alicante, Alicante
  - Hospital General Universitario de Elche, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Universitari de Bellvitge, Barcelona
  - IrsiCaixa, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
- United Kingdom (8):
  - Elton John Centre, Brighton
  - Southmead Hospital, Bristol
  - Bart's Hospital, London
  - Royal Free Hospital, London
  - St Thomas Hospital, London
  - Chelsea & Westminster Hospital, London
  - St Mary's Hospital, London
  - Mortimer Market Centre, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Waters L, Assoumou L, Gonzalez-Cordon A, Rusconi S, Domingo P, Gompels M, de Wit S, Raffi F, Stephan C, Masia M, Rockstroh J, Katlama C, Behrens GMN, Moyle G, Johnson M, Fox J, Stellbrink HJ, Guaraldi G, Florence E, Esser S, Gatell JM, Pozniak A, Martinez E; NEAT 022 Study Group. Limited Weight Impact After Switching From Boosted Protease Inhibitors to Dolutegravir in Persons With Human Immunodeficiency Virus With High Cardiovascular Risk: A Post Hoc Analysis of the 96-Week NEAT-022 Randomized Trial. Clin Infect Dis. 2023 Mar 4;76(5):861-870. doi: 10.1093/cid/ciac827. PMID 36259527
- [Derived] Saumoy M, Sanchez-Quesada JL, Assoumou L, Gatell JM, Gonzalez-Cordon A, Guaraldi G, Domingo P, Giacomelli A, Connault J, Katlama C, Masia M, Ordonez-Llanos J, Pozniak A, Martinez E, Podzamczer D. Atherogenicity of low-density lipoproteins after switching from a protease inhibitor to dolutegravir: a substudy of the NEAT022 study. J Antimicrob Chemother. 2022 Jun 29;77(7):1980-1988. doi: 10.1093/jac/dkac117. PMID 35411401
- [Derived] Gatell JM, Assoumou L, Moyle G, Waters L, Johnson M, Domingo P, Fox J, Martinez E, Stellbrink HJ, Guaraldi G, Masia M, Gompels M, De Wit S, Florence E, Esser S, Raffi F, Stephan C, Rockstroh J, Giacomelli A, Vera J, Bernardino JI, Winston A, Saumoy M, Gras J, Katlama C, Pozniak AL; European Network for AIDS Treatment 022 (NEAT022) Study Group. Immediate Versus Deferred Switching From a Boosted Protease Inhibitor-based Regimen to a Dolutegravir-based Regimen in Virologically Suppressed Patients With High Cardiovascular Risk or Age >/=50 Years: Final 96-Week Results of the NEAT022 Study. Clin Infect Dis. 2019 Feb 1;68(4):597-606. doi: 10.1093/cid/ciy505. PMID 29912307